CLINICAL TRIAL: NCT04768491
Title: Real-world Study on Sequential Therapy With Dacomitinib as First-line Treatment Followed by 3rd Generation EGFR-TKI in Patients With EGFR Mutation Positive Advanced Non-Small Cell Lung Cancer
Brief Title: Dacomitinib Treatment Followed by 3rd Generation EGFR-TKI in Patients With EGFR Mutation Positive Advanced NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Junling Li, professor, Peking Union Medical College
Other Study IDs: NCC2439
Record Dates: First submitted 2021-02-18; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: EGFR Activating Mutation; NSCLC Stage IV; NSCLC Stage IIIB; NSCLC, Recurrent
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence | interventions — dacomitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample will be taken when each patient were reexamined in hospital
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- dacomitinib treatment: Sequential Therapy with Dacomitinib as First-line Treatment Followed by 3rd generation EGFR-TKI in Patients with EGFR Mutation Positive Advanced Non-Small Cell Lung Cancer
  Interventions: Drug: Dacomitinib

INTERVENTIONS:
Drug: Dacomitinib — effectiveness and safety profile in patients with EGFR mutation-positive advanced NSCLC treated with dacomitinib (Vizimpro®) as the first-line treatment followed by 3rd generation EGFR-TKI in case the T790M resistance mutation was developed.

SUMMARY:
This is a non-interventional, multi-center, ambispective cohort study in real world to describe the effectiveness and safety profile in patients with EGFR mutation-positive advanced NSCLC treated with dacomitinib (Vizimpro®) as the first-line treatment followed by 3rd generation EGFR-TKI in case the T790M resistance mutation was developed.

DETAILED DESCRIPTION:
This is a multi-center observational study with both retrospective and prospective data collections to describe the effectiveness and safety of sequential dacomitinib and 3rd generation EGFR-TKI used in patients with EGFR mutation-positive NSCLC with T790M-aquired resistance in a clinical practice setting. The study will include patients who were or will be diagnosed as advanced NSCLC with EGFR mutation positive and received dacomitinib as first-line treatment followed by second-line 3rd generation EGFR-TKI treatment in multiple tertiary care hospitals after Sep 1st, 2019. Patients' clinical information prior to the study initiation in each hospital will be collected retrospectively through chart review. After the study initiation, new patient enrollment will last till Dec 2022. Patients' clinical care after the study initiation will be followed up prospectively until the end of study. The interval of response evaluation is recommended to be every 2 to 3 months in the treatment period and the interval of follow-up is recommended to be every 2 to 3 months in the post-treatment period till the end of study in the prospective data collection period.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of locally advanced or metastatic NSCLC.
* The tumor harbored common EGFR mutations (Del19, L858R) at start of first-line treatment
* Age ≥ 18 years
* Had never received any EGFR TKI therapy.
* Patients that treated with dacomitinib (Vizimpro®) as first-line treatment
* Confirmation of the T790M variant after first line dacomitinib treatment and receive any 3rd generation EGFR-TKI as second-line treatment.
* Asymptomatic CNS metastases allowed
* At least one lesion that can be accurately measured at baseline according to the RECIST 1.1, and which is suitable for accurate repeated measurements.
* Start second-line treatment with third generation EGFR TKI no later than 01 JAN2023（>10 month before data cutoff date）
* All eligible patients are required to sign an informed consent before initiating the study

Exclusion Criteria:

* Patients who received drug(s) other than 3rd generation EGFR-TKI as the second-line treatment and/or patients who received drug(s) other than Dacomitinib (Vizimpro®) as the first-line treatment
* Received or currently receiving dacomitinib from any interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with EGFR mutation and advanced NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
time to treatment failure | up to 4 years
  To describe the time to treatment failure (TTF) of sequential dacomitinib and 3rd generation EGFR-TKI used in patients with EGFR mutation-positive NSCLC and T790M-aquired resistance in China.

SECONDARY OUTCOMES:
progression-free survival | up to 4 years
  To describe the progression-free survival (PFS) of dacomitinib and 3rd generation EGFR-TKI used in patients with EGFR mutation-positive NSCLC with T790M-aquired resistance in China.
duration of treatment | up to 4 years
  To describe the duration of treatment (DOT) of dacomitinib and 3rd generation EGFR-TKI used in patients with EGFR mutation-positive NSCLC with T790M-aquired resistance respectively in China.
overall survival | up to 5 years
  To describe the overall survival (OS) of sequential dacomitinib and 3rd generation EGFR-TKI used in patients with EGFR mutation-positive NSCLC and T790M-aquired resistance in China.

CONTACTS AND LOCATIONS:
Overall Officials: Junling Li, MD, Study Director — Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No